CLINICAL TRIAL: NCT01660308
Title: Observing the Changes of Fibroblast Growth Factor 23 in Patients of Tumor Induced Osteomalacia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201105045RC
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tumor induced osteomalcia

SUMMARY:
Fibroblast froth factors (FGFs) are humoral factors identified by their ability to stimulate cell proliferation1. They play different roles in the regulation of cell proliferation, differentiation and function. Most FGF family members act as paracrine factors. But FGF19(FGF19) subfamily members, including FGF19, 21, and 23, work as endocrine factors to regulate bile acid, carbohydrate and phosphate metabolism2. Of these, FGF23 plays an important role in phosphate and bone metabolism3. FGF23 gene encodes 251 amino acids, including a 24-amino acid signal peptide4. The secreted FGF23 is a protein consisted of 227 amino acids. It works by binding to a Klotho-FGF receptor 1c (FGF1c) complex5. FGF suppresses the expression of type 2a and 2c sodium-phosphate cotransporters, which mediate phosphate reabsorption in proximal tubules.6 FGF23 decreases 25-hydroxyvitamin D-1α-hydroxylase expression and enhances 25-hydroxyvitamin D-24-hydroxylase expression6. Therefore, FGF23 reduces serum 1,25-dihydroxyvitamin D〔1,25(OH)2D〕, which stimulates intestinal calcium and phosphate absorption. FGF23 decreases serum phosphate through the above mechanisms FGF23 over-expression might result in hypophosphatemic rickets and osteomalacia.

Tumor induced osteomalacia (TIO) is a paraneoplastic syndrome usually caused by benign phosphaturic mesenchymal tumors. Symptoms are nonspecific, such as general weakness, fatigue, and bone pain. Sometimes fracture may occurs. The responsible tumors are sometimes small and difficult to detect. Tumors secrete FGF23. FGF23 reduced phosphate reabsorption in the proximal tubules and decrease 1,25(OH)2D levels, which result in hypophosphatemia and then osteomalacia.

The investigators would like to observe the changes of FGF23 in patients who receive operation or medical treatment and hope this will benefit future treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with tumor induced osteomalacia.
* people without osteomalacia such as healthy people,
* people under dialysis,
* people with poor nutrition.

Exclusion Criteria:

* people younger than 20 years old or older than 85 years old.
* people who are pregnant.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with tumor induced osteomalacia and people without osteomalacia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
FGF23, P | at the time TIO is diagnosed

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Lin CH, Chang CK, Shih CW, Li HY, Chen KY, Yang WS, Tsai KS, Wang CY, Shih SR. Serum fibroblast growth factor 23 and mineral metabolism in patients with euthyroid Graves' diseases: a case-control study. Osteoporos Int. 2019 Nov;30(11):2289-2297. doi: 10.1007/s00198-019-05116-1. Epub 2019 Aug 5. PMID 31384956
- [Derived] Lin HA, Shih SR, Tseng YT, Chen CH, Chiu WY, Hsu CY, Tsai KS. Ovarian cancer-related hypophosphatemic osteomalacia--a case report. J Clin Endocrinol Metab. 2014 Dec;99(12):4403-7. doi: 10.1210/jc.2014-2120. PMID 25181387